CLINICAL TRIAL: NCT06865638
Title: A Comparative Study of Clinical Outcomes Between Leak Testing and No Leak Testing for Anastomosis in Colorectal Cancer Surgery: a Multicenter, Stratified Randomized Controlled Trial.
Brief Title: Efficacy and Safety of Colorectal Anastomotic Leak Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025008
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Leakage Testing; Colorectal Surgery; Complications; Anastomotic Leakage
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- ≤5cm Rectal, Pre-chemo, Leak Test (Experimental): Patients with rectal cancer ≤ 5 cm from the anus, received preoperative chemotherapy and intraoperative leak testing.
  Interventions: Procedure: Intraoperative leak testing
- ≤5cm Rectal, Pre-chemo, No Leak Test (No Intervention): Patients with rectal cancer ≤ 5 cm from the anus, received preoperative chemotherapy, and had no intraoperative leak testing.
- ≤5cm Rectal, No pre-chemo, Leak Test (Experimental): Patients with rectal cancer ≤ 5 cm from the anus, didn't receive preoperative chemotherapy, and underwent intraoperative leak testing.
  Interventions: Procedure: Intraoperative leak testing
- ≤5cm Rectal, No pre-chemo, No Leak Test (No Intervention): Patients with rectal cancer ≤ 5 cm from the anus, didn't receive preoperative chemotherapy, and had no intraoperative leak testing.
- >5cm Colorectal, Pre-chemo, Leak Test (Experimental): Patients with colorectal cancer > 5 cm from the anus, received preoperative chemotherapy, and underwent intraoperative leak testing.
  Interventions: Procedure: Intraoperative leak testing
- >5cm Colorectal, Pre-chemo, No Leak Test (No Intervention): Patients with colorectal cancer > 5 cm from the anus, received preoperative chemotherapy, and had no intraoperative leak testing.
- >5cm Colorectal, No pre-chemo, Leak Test (Experimental): Patients with colorectal cancer > 5 cm from the anus, didn't receive preoperative chemotherapy, and underwent intraoperative leak testing.
  Interventions: Procedure: Intraoperative leak testing
- >5cm Colorectal, No pre-chemo, No Leak Test (No Intervention): Patients with colorectal cancer > 5 cm from the anus, didn't receive preoperative chemotherapy, and had no intraoperative leak testing.

INTERVENTIONS:
Procedure: Intraoperative leak testing — ◦After anastomosis was completed, the integrity of anastomosis was tested intraoperatively. The methods include directly observing the integrity of the anastomosis under gastroscopy, immersing the anastomosis in 500 - 1000 mL of warm saline and temporarily occluding the distal end, filling the anastomotic bowel with air, and injecting 60 mL of methylene blue through colonoscopy. Wrapping a white gauze pad around the anastomosis and observing for methylene blue leakage.
  Arms: >5cm Colorectal, No pre-chemo, Leak Test; >5cm Colorectal, Pre-chemo, Leak Test; ≤5cm Rectal, No pre-chemo, Leak Test; ≤5cm Rectal, Pre-chemo, Leak Test

SUMMARY:
To evaluate the effectiveness of the gastroscopy, air, and methylene blue (GAM) leak testing in reducing the incidence of postoperative anastomotic complications, especially anastomotic leakage, in patients with colorectal cancer. The primary outcomes included is the incidence of anastomotic complications (mainly anastomotic leak) within 30 days after surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with colorectal cancer by pathology and scheduled for surgical treatment who meet the surgical indications.
2. Aged between 18 and 85 years.
3. American Society of Anesthesiologists (ASA) physical status classification is I - III.
4. The patient or his/her legal representative can understand and sign the informed consent form and is willing to cooperate throughout the study process.

Exclusion Criteria:

1. Patients with preoperatively diagnosed anastomotic leak or other severe abdominal infections.
2. Patients with severe cardiovascular and cerebrovascular diseases (such as recent myocardial infarction, unstable angina pectoris, severe heart failure, acute cerebral infarction, etc.) who cannot tolerate surgery and related tests.
3. Patients with severely impaired liver and kidney function (liver function Child - Pugh classification C or above, creatinine clearance rate < 30 ml/min).
4. Patients with coagulation disorders (such as platelet count < 50×10⁹/L, international normalized ratio (INR) > 1.5, etc.) that cannot be corrected or are receiving anticoagulant therapy that cannot be adjusted.
5. Patients with a history of abdominal radiotherapy or multiple abdominal surgeries and severe abdominal adhesions that may affect the operation and detection procedures.
6. Patients with other malignant tumors who are receiving active anti-tumor treatment such as radiotherapy and chemotherapy.
7. Patients with mental illness or cognitive impairment who cannot cooperate with the study process and follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Anastomotic Leak within 30 days | 30 days
  Count the number of participants who develop anastomotic leak within 30 days after colorectal cancer surgery.

SECONDARY OUTCOMES:
Number of Participants with Postoperative Complications within 30 days | 30 days
  Count the number of participants who develop postoperative bleeding, anastomotic stenosis, and intra-abdominal infection within 30 days after colorectal cancer surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China